CLINICAL TRIAL: NCT01327300
Title: Randomized, Double-blind, Cross-over Study of the Efficacy of Mesalamine in Diarrhea-predominant Irritable Bowel Syndrome (dIBS)
Brief Title: Efficacy of Mesalamine in Diarrhea-predominant Irritable Bowel Syndrome (dIBS)
Acronym: IBS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 106-2010
Record Dates: First submitted 2011-03-24; First posted 2011-04-01 (Estimated); Results first posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Irritable Bowel Syndrome Treatment; Mesalamine; Anti-inflammatory drugs; 5-ASA drugs; Apriso ™
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mesalamine (Active Comparator): This group received the drug Mesalamine for 12 weeks then a wash out for 3 weeks prior to crossing over to the placebo arm.
  Interventions: Drug: Mesalamine
- Placebo (Placebo Comparator): This group will receive the Placebo for 12 weeks then a wash out for 3 weeks prior to crossing over to the drug arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mesalamine — Apriso is a 5-ASA drug with Intellicor ™ extended-release delivery technology. A 1.5 gram dosage of Apriso (equaling four 375 mg capsules) once a day will be administered orally for a period of 12 weeks followed by a 3 week wash out prior to crossing over to the placebo arm.
  Other Names: Apriso ™
  Arms: Mesalamine
Other: Placebo — 4 capsules (.375 gm sugar pill capsules) administered orally once a day. This group will receive the placebo for 12 weeks then a wash out for 3 weeks prior to crossing over to the drug arm.
  Arms: Placebo

SUMMARY:
The purpose of this study is to find whether treating patients with diarrhea predominant Irritable Bowel Syndrome (IBS) with an anti-inflammatory drug called Mesalamine will help improve their symptoms of diarrhea, bloating and abdominal pain.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a common gastrointestinal disorder affecting about 20% of the United States population and comprising almost 50% of referrals to gastroenterology practices. Although the pathophysiology of IBS is poorly understood, more recently, both inflammation and an increased intestinal permeability have been identified as potential factors in the etiology of diarrhea-predominant IBS patients(dIBS). Despite the potential of an inflammatory etiology for IBS, few studies have examined the efficacy of anti-inflammatory agents such as mesalamine in patients with IBS. The primary objective of our study is to determine the efficacy of Apriso™ (Salix Pharmaceuticals Inc), a long-acting mesalamine, in the treatment of patients with dIBS. Apriso™, is a mesalamine approved by the Food and Drug Administration (FDA) on October 31, 2008 for the maintenance of remission in patients with active, mild to moderate ulcerative colitis. The investigators will perform a randomized, double-blind, cross-over trial of mesalamine compared to placebo in patients with dIBS. This study will analyze both the objective and subjective measures of improvement in IBS symptoms. The subjective measures will include improvements in the overall symptom severity scores and the Global Improvement Scale (GIS) and the objective measures will include histological measures of inflammation as well as improvements in the intestinal membrane permeability of treated subjects. The investigators will demonstrate that during the 12 weeks treatment period with mesalamine, subjects will have improvements in their overall symptom scores, GIS scores, and will have a reduction in intestinal inflammation and also prohibit a likely improvement in Intestinal membrane permeability.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 18-65 years old
* Functional Bowel Disorder Severity Index Score above 37
* Normal complete blood count, liver function studies and renal function studies
* Serologies done to rule out Celiac Spure or patient has prior negative EGD with small bowel biopsies which have been negative
* Infectious diarrhea ruled out by stool studies
* Negative colonoscopy

Exclusion Criteria:

* Any history of chronic liver disease, heart disease, pulmonary or renal disease
* Abnormal EKG
* Women with positive pregnancy tests
* Patient on steroids, antacids, or warfarin or chronic pain conditions other than fibromyalgia
* Patients who drink over 2oz alcohol/day on a regular basis Any other causes for diarrhea such as IBD, microscopic colitis, celiac disease, history of abdominal obstruction, pancreatitis, ileus, or any gastrointestinal bleeding.
* Patients with active malignancy in the past five years
* Patient with any history of hypersensitivity reactions to salicylate containing medications due to cross-sensitivity with mesalamine or allergy to mesalamine medications in the past
* Any subjects with fibromyalgia will be excluded from the pain testing portion only
* History of Phenylketonuria due to the aspartame contained in Apriso

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baharak Moshiree, MD, MS, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Drossman DA, Whitehead WE, Camilleri M. Irritable bowel syndrome: a technical review for practice guideline development. Gastroenterology. 1997 Jun;112(6):2120-37. doi: 10.1053/gast.1997.v112.agast972120. No abstract available. PMID 9178709
- [Background] Sandler RS. Epidemiology of irritable bowel syndrome in the United States. Gastroenterology. 1990 Aug;99(2):409-15. doi: 10.1016/0016-5085(90)91023-y. PMID 2365191
- [Background] Bjarnason I, MacPherson A, Hollander D. Intestinal permeability: an overview. Gastroenterology. 1995 May;108(5):1566-81. doi: 10.1016/0016-5085(95)90708-4. PMID 7729650
- [Background] Dunlop SP, Hebden J, Campbell E, Naesdal J, Olbe L, Perkins AC, Spiller RC. Abnormal intestinal permeability in subgroups of diarrhea-predominant irritable bowel syndromes. Am J Gastroenterol. 2006 Jun;101(6):1288-94. doi: 10.1111/j.1572-0241.2006.00672.x. PMID 16771951
- [Background] Corinaldesi R, Stanghellini V, Cremon C, Gargano L, Cogliandro RF, De Giorgio R, Bartesaghi G, Canovi B, Barbara G. Effect of mesalazine on mucosal immune biomarkers in irritable bowel syndrome: a randomized controlled proof-of-concept study. Aliment Pharmacol Ther. 2009 Aug;30(3):245-52. doi: 10.1111/j.1365-2036.2009.04041.x. Epub 2009 May 12. PMID 19438846
- [Background] Gordon S, Ameen V, Bagby B, Shahan B, Jhingran P, Carter E. Validation of irritable bowel syndrome Global Improvement Scale: an integrated symptom end point for assessing treatment efficacy. Dig Dis Sci. 2003 Jul;48(7):1317-23. doi: 10.1023/a:1024159226274. PMID 12870789
- [Background] Zhou Q, Fillingim RB, Riley JL 3rd, Malarkey WB, Verne NG. Central and peripheral hypersensitivity in the irritable bowel syndrome. Pain. 2010 Mar;148(3):454-461. doi: 10.1016/j.pain.2009.12.005. Epub 2010 Jan 13. PMID 20074857
- [Background] Myers CD, Robinson ME, Riley JL 3rd, Sheffield D. Sex, gender, and blood pressure: contributions to experimental pain report. Psychosom Med. 2001 Jul-Aug;63(4):545-50. doi: 10.1097/00006842-200107000-00004. PMID 11485107

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the gastroenterology specialty clinics at the University of Florida or by referral from other primary care physicians. Recruitment was from 2011 until March, 2012
Pre-assignment Details: A washout period of 3 weeks was given between treatment periods with 2 weeks prior to recruitment.
Groups:
- Mesalamine Then Placebo: This group received the drug Mesalamine for 12 weeks then a wash out for 3 weeks prior to crossing over to the placebo arm.
  Mesalamine : Apriso is a 5-ASA drug with Intellicor ™ extended-release delivery technology. A 1.5 gram dosage of Apriso (equaling four 375 mg capsules) once a day will be administered orally for a period of 12 weeks followed by a 3 week wash out prior to crossing over to the placebo arm.
- Placebo Then Mesalamine: This group will receive the Placebo for 12 weeks then a wash out for 3 weeks prior to crossing over to the drug arm.
  Placebo : 4 capsules (.375 gm sugar pill capsules) administered orally once a day. This group will receive the placebo for 12 weeks then a wash out for 3 weeks prior to crossing over to the drug arm.
Period: First Intervention (12 Weeks)
Arm/Group | Mesalamine Then Placebo | Placebo Then Mesalamine
Started | 5 | 2
Completed | 5 | 2
Not Completed | 0 | 0
Period: Washout (3 Weeks)
Arm/Group | Mesalamine Then Placebo | Placebo Then Mesalamine
Started | 5 | 2
Completed | 4 | 2
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention (12 Weeks)
Arm/Group | Mesalamine Then Placebo | Placebo Then Mesalamine
Started | 4 | 2
Completed | 4 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants were randomized to receive both mesalamine and placebo.
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Changes in GIS Scores Between Baseline and After a 12 Week Intervention With Mesalamine or Placebo
Description: Patients rated the severity of their GI symptoms. The GIS scale goes from 1 to 7 with 1 being the worse and 7 as the best score showing improvement in symptoms. The GIS was performed at week one and at week 12 during each of the interventions. The comparisons below list the mean difference for each intervention from baseline (BL) with standard deviations then we list the p-value for the differences of baseline to intervention are reported using the Mann-Whitney test with a two-tailed p value provided.
Time Frame: Baseline and at 12 weeks post-intervention
Population: The first part of the analysis compares the differences between baseline and mesalamine to baseline and placebo. The P value provided below list the comparison of baseline-placebo to baseline-mesalamine using the Mann-Whitney statistical analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mesalamine: This group received the drug Mesalamine for 12 weeks Mesalamine : Apriso is a 5-ASA drug with Intellicor ™ extended-release delivery technology. A 1.5 gram dosage of Apriso (equaling four 375 mg capsules) once a day will be administered orally for a period of 12 weeks
- Placebo: This group will receive the Placebo for 12 weeks.
  Placebo : 4 capsules (.375 gm sugar pill capsules) administered orally once a day. This group will receive the placebo for 12 weeks.
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 7 | 6
units on a scale | 2.72 (1.82) [4.52 to 5.14] | 2.22 (1.49) [2.24 to 3.18]
Statistical Analysis 1: Comparison: Mesalamine; The GIS scoring system is from 1-7 with one being a worse outcome and 7 the better outcome. Comparisons below list the p values for comparison of difference in GIS between baseline and mesalamine; Test type: Superiority or Other; p = .001, t-test, 2 sided; Mean Difference (Final Values) = 2.72
Statistical Analysis 2: Comparison: Placebo; Comparisons of mean difference in GIS scores between baseline and placebo is made below; Test type: Superiority or Other; p = 0.008, t-test, 2 sided; Mean Difference (Final Values) = 2.22

2. Secondary Outcome: Number of Participants Who Had Evidence of Increased Levels of Pathologic Indicators of Colonic Mucosal Inflammation at 12 Weeks Compared to Baseline.
Description: Colonoscopy/flexible sigmoidoscopy will be performed and mucosal biopsies will be obtained. Each biopsy was stained for activated t lymphocytes, mast cells and eosinophils .
  CD117 staining was done for Mast cells. H and E staining was used to identify lymphocytes and eosinophils. Each path specimen was then noted to have increased versus normal number of these inflammatory cells.
Time Frame: For 2 times: First time: at the time of patient recruitment in the study Second time: after the completion of first 12-week treatment period, all of which are during the time period from 02/25/2010 to 02/01/2012 (up to 2 years)
Measure: Number; unit: participants
Groups:
- Mesalamine: This group received the drug Mesalamine for 12 weeks then a wash out for 3 weeks prior to crossing over to the placebo arm.
  The data below reflect the change in the increase in inflammation with regards to increased mast cells, eosinophils counts and number of activated T lymphocytes after 12 week mesalamine from baseline level of inflammation.
- Placebo: This group will receive the Placebo for 12 weeks then a wash out for 3 weeks prior to crossing over to the drug arm.
  The data below reflect the change in the increase in inflammation with regards to increased mast cells, eosinophils counts and number of activated T lymphocytes after 12 week mesalamine from baseline level of inflammation
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 7 | 6
participants
  Increased Mast cells-CD 117 Positive staining | 2 | 2
  Increased eosinophil counts | 3 | 3
  Increased Activated T lymphocytes-CD3 | 2 | 3
Statistical Analysis 1: Comparison: Mesalamine; Correlation coefficients were used for each of three biomarkers in relation to other biomarkers and to the questionnaires and patient's symptoms; Test type: Superiority or Other; p = 0.873, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; The study tested three biomarkers and symptom domains at baseline and the end of 12 weeks of placebo using the Mann-Whitney test, as well as correlations between domains with Pearson's linear correlation coefficient; Test type: Superiority or Other; p = 0.810, Wilcoxon (Mann-Whitney); Pearson's linear coefficient

3. Secondary Outcome: Functional Bowel Disorder Severity Index (FBDSI)
Description: Subjects rate pain on a standardized scale. This is a standardized test used to evaluate patients with IBS. Baseline values are compared to 12 weeks after mesalamine and 12 weeks after placebo treatments. The FBDSI is score is interpreted as such: Severity of IBS is rated as none (0 points), mild (1-36 points), moderate as 37-110 points and severe as >110 points. Therefore patients can have a score higher than 110.
Time Frame: An FBDSI score is administered at the beginning of each 12-week treatment period (baseline) and at the end of each 12-week treatment period.
Population: Change in Functional Bowel Disorder Severity Index (FBDSI)after 12 weeks of intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mesalamine: This group received the drug Mesalamine for 12 weeks then a wash out for 3 weeks prior to crossing over to the placebo arm.
  Data is reported as baseline value minus 12 week mean FBDSI value with mesalamine.
- Placebo: This group will receive the Placebo for 12 weeks then a wash out for 3 weeks prior to crossing over to the drug arm.
  Values reported at the baseline FBDSI score minus the 12 week FBDSI score with placebo.
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 7 | 6
units on a scale | -14.5 (61.5) [0 to 197] | 17 (71) [0 to 209]
Statistical Analysis 1: Comparison: Mesalamine; The FBDSI score is based on the severity of abdominal pian. Severity is rated as the following: None= 0 points Mild= (1-36) Moderate =(37-110) Severe= (>110 points); Test type: Superiority or Other; p = 0.67, t-test, 2 sided; Two-tailed P values are listed for baseline versus 12 weeks of mesalamine; Mean Difference (Final Values) = -14.5
Statistical Analysis 2: Comparison: Placebo; See prior description of the FBDSI score. Change in the FBDSI after 12 weeks of intervention is made using a two sided t-test; Test type: Superiority or Other; p = 0.77, t-test, 2 sided; Mean Difference (Final Values) = 17

4. Secondary Outcome: IBS - Quality of Life (IBS-QOL)Score.
Description: A questionnaire is given to each patient and was completed at baseline then after 12 weeks of intervention with mesalamine and then placebo in the cross-over study. The IBS-QOL comprises 34 items with 5-point response scales (0 to 4) that cover eight dimensions of HRQL: dysphoria (8 items), interference with activity (7 items), body image (4 items), health worry (3 items),food avoidance (3 items), social reaction (4 items), sexual concerns (2 items) and relationships (3 items). Higher values indicate better HRQL after converting the raw score on the IBS-QOL into 0 to 100 points.
Time Frame: at the time of recruitment and after completion of each 12-week treatment period, all of which are during the time period from 03/25/2010 to 02/01/2012 (up to 2 years)
Population: Data are the mean change in IBS-QOL between baseline and intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mesalamine: This group received the drug Mesalamine for 12 weeks.
  The data below show the change in IBS-QOL scores from baseline after 12 weeks of intervention.
- Placebo: This group will receive the Placebo for 12 weeks.
  The data below show the change in IBS-QOL scores from baseline after 12 weeks of intervention.
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 7 | 6
units on a scale | 11 (36.1) [40 to 163] | -12.2 (28.2) [38 to 124]
Statistical Analysis 1: Comparison: Mesalamine; For the IBS QOL we compared the change in IBS-Quality of Life (IBS-QOL) after 12 weeks of mesalamine; Test type: Superiority or Other; p = 0.61, t-test, 2 sided; Mean Difference (Final Values) = 11
Statistical Analysis 2: Comparison: Placebo; Comparison of change in IBS-Quality of Life (IBS-QOL)from baseline after 12 weeks of intervention was made; Test type: Superiority or Other; p = 0.33, t-test, 2 sided; Mean Difference (Final Values) = -12.2

5. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS)
Description: A questionnaire is given to each patient with scoring done on a Likert scale ranking from 0-42 which combines anxiety and depression scales. Each of these are scored from 0-21 depending on anxiety versus the depression parameters. Comparison of change in HADs after 12 weeks of intervention with either mesalamine or placebo is provided here with only the total value provided-range is from 0-42.
  Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 3 with zero being none at all or occasional and 3 as most of the time. The scale used is a Likert scale and therefore the data returned from the HADS is ordinal.
  The best score for the HADS therefore is a 0 with the worst score a 42 for combined anxiety and depression scores.
  For the subscales of depression and anxiety, the best score is a 0 and the worst is a 21. This data is not provided here.
  Data below includes the change from baseline in the HADS scores.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mesalamine: This group received the drug Mesalamine for 12 weeks . Comparison of the change in HADS score after 12 weeks of mesalamine is made to baseline score.
- Placebo: This group will receive the Placebo for 12 weeks. Comparison of the change in HADS score after 12 weeks of placebo is made to baseline score.
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 7 | 6
units on a scale
  HADS score- change from baseline c/w 12 weeks | 1.2 (6.1) | -2.4 (8.7)
  HADS Score-end of 12 weeks | 14 (6.3) | 13 (10.3)
Statistical Analysis 1: Comparison: Mesalamine; Comparison of the change in HADS score of baseline to 12 weeks of mesalamine is made; Test type: Superiority or Other; p = 0.71, t-test, 2 sided; Mean Difference (Final Values) = 1.3
Statistical Analysis 2: Comparison: Placebo; Comparison of change in HADS score between baseline and after 12 weeks of placebo is made; Test type: Superiority or Other; p = 0.57, t-test, 2 sided; Mean Difference (Final Values) = -2.4

6. Secondary Outcome: Intestinal Permeability Testing
Description: Ability of test substances to permeate the intestinal mucosa. The Lactulose/Mannitol test (Genova Diagnostics®, Ashville, NC) directly measures the ability of mannitol and lactulose to permeate the intestinal mucosa. Patient ingests 5 grams of lactulose and 2 grams of mannitol dissolved in a 100 ml of water. Urine is then collected for 24 hours and the ratio of the urinary excretion of lactulose to mannitol is measured. This testing is performed only after completion of each treatment period , after 12 weeks of mesalamine and after 12 weeks of placebo.
  Normal ratio of lactulose/mannitol is any value <0.7. An abnormal ratio is defined as >0.7 ratio. The lactulose is measured in the urine as g/kg and the urinary excretion of mannitol is also measures as g/kg.
Time Frame: At the completion of each 12-week treatment period, all of which are during the time period from 03/25/2010 to 02/01/2012 (up to 2 years)
Measure: Mean (Full Range); unit: ratio
Groups:
- Mesalamine: This group received the drug Mesalamine for 12 weeks and after a 12 week treatment period, the ratio of lactulose to mannitol was measured.
- Placebo: This group received the placebo for 12 weeks and after a 12 week treatment period, the ratio of lactulose to mannitol was measured.
  Two patients in this cross-over study did not provide a 24 hour urine sample needed to obtain the lactulose /mannitol ratio.
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 7 | 5
ratio | 0.07 [0.03 to 0.11] | 0.04 [0.02 to 0.05]
Statistical Analysis 1: Comparison: Mesalamine vs Placebo; Comparison of the lactulose/mannitol ratio is made after a 12 week intervention with mesalamine to 12 weeks of placebo; Test type: Superiority or Other; p = 0.55, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Mesalamine Then Placebo | Placebo Then Mesalamine
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 0/5 | 0/2

LIMITATIONS AND CAVEATS:
The recruitment for this study ended on 3/2012 when Dr. Moshiree became adjunct faculty only at the University Florida. This study was limited with over 6 months of follow-up and the need for three endoscopies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No